CLINICAL TRIAL: NCT04333147
Title: A Multi-centre Long-term Extension Study to Assess the Safety and Efficacy of GSK3196165 in the Treatment of Rheumatoid Arthritis
Brief Title: Long-term Safety and Efficacy of GSK3196165 (Otilimab) in the Treatment of Rheumatoid Arthritis (RA)
Acronym: contRAst X
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study is early terminated due to Limited efficacy demonstrated in the contRAst program does not support a suitable benefit/risk profile for otilimab as a potential treatment for RA. GSK has decided not to progress with regulatory submissions.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 209564
Record Dates: First submitted 2020-03-27; First posted 2020-04-03 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; GSK3196165; Otilimab; Long-term safety; Long-term efficacy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab

STUDY DESIGN:
Intervention Model Description: Participants who received GSK3196165 in their qualifying study will continue in this study on the same dose. Participants who received a comparator (tofacitinib or sarilumab) in their qualifying study will be centrally randomized using interactive response technology (IRT) in a ratio of 1:1 to either GSK3196165 90 mg or 150 mg.
Who Masked: Participant, Investigator
Masking Description: This is a parallel group treatment study with two arms that are initially participant and investigator blinded. A participant's treatment allocation will remain blinded at least until their qualifying study has been reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Otilimab 90 mg (Experimental): Participants who received Otilimab 90mg in a qualifying study and continued on Otilimab 90mg in study 209564 or participants who received either tofacitinib 5mg (study 201790 or 201791) or sarilumab 200mg (study 202018) in a qualifying study and were exposed for the first time to Otilimab 90mg in study 209564. Otilimab 90mg was administered through subcutaneous (SC) injection once weekly.
  Interventions: Biological: Otilimab (GSK3196165); Drug: csDMARD(s)
- Otilimab 150 mg (Experimental): Participants who received Otilimab 150mg in a qualifying study and continued on Otilimab 150mg in study 209564 or participants who received either tofacitinib 5mg (study 201790 or 201791) or sarilumab 200mg (study 202018) in a qualifying study and were exposed for the first time to Otilimab 150mg in study 209564. Otilimab 150mg was administered through subcutaneous (SC) injection once weekly.
  Interventions: Biological: Otilimab (GSK3196165); Drug: csDMARD(s)

INTERVENTIONS:
Biological: Otilimab (GSK3196165) — GSK3196165 solution in vial/pre-filled syringe (PFS) and auto injector (AI) to be administered SC.
Drug: csDMARD(s) — Stable dose of csDMARD(s) as standard of care (SoC).

SUMMARY:
RA is a chronic, systemic inflammatory autoimmune disease which requires treatment for a long time period, hence it is important to study the long-term safety and efficacy of the continuous treatment with GSK3196165 over several years. This is a Phase 3, multicenter, parallel group treatment and long-term extension study primarily to assess safety with efficacy assessment as a secondary objective. Adult participants with RA who have completed the treatment phase of a qualifying GSK3196165 clinical studies (Phase 3 studies contRAst 1 (201790: NCT03980483), contRAst 2 (201791: NCT03970837) and contRAst 3 (202018: NCT04134728) and who, in investigator's judgement will benefit from extended treatment with GSK3196165 will be included in this study (contRAst X [209564: NCT04333147]). Participants will continue to receive the same background conventional synthetic disease modifying anti-rheumatic drug(s) [csDMARD(s)] treatment as they received in their qualifying study. Eligible participants will be enrolled to receive weekly GSK3196165 90 milligrams (mg) or 150 mg by subcutaneous (SC) injection. The anticipated study duration is approximately 4 years which will enable participants to receive treatment with GSK3196165 until it is expected to become commercially available. Approximately 3000 participants from the qualifying studies will participate in this long-term extension study

ELIGIBILITY:
Inclusion Criteria:

* Participants with rheumatoid arthritis who are aged >=18 years at the time of signing informed consent, who have completed one of the qualifying GSK3196165 clinical studies and who, in the opinion of the investigator, may benefit from treatment with GSK3196165.
* Body weight >=40 kilograms (kg).
* Male or female participants are eligible to participate as long as they meet the contraceptive eligibility criteria and agree to abide by the contraceptive requirements.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* For participants on methotrexate (MTX): must be willing to continue treatment with oral folic acid (at least 5 mg/week) or equivalent while receiving MTX (mandatory co-medication for MTX treatment).

Exclusion Criteria:

* Had study intervention permanently discontinued at any time during a qualifying study except any participant with a new diagnosis of latent Mycobacterium tuberculosis (TB) at the end of study assessment in a qualifying study and currently undertaking or willing to complete at least 4 weeks of anti-TB treatment off study treatment, per world health organization (WHO) or national guidelines prior to re-commencing therapy and complete the remainder of anti-TB treatment while on study.
* Evidence of latent TB (as documented by a positive QuantiFERON-TB Gold plus test or T-SPOT.TB test, no findings on medical history or clinical examination consistent with active TB, and a normal chest radiograph) except for participants that

  * Are currently undertaking or willing to complete at least 4 weeks of anti-TB therapy off study treatment, as per WHO or national guidelines prior to re- commencing study treatment and agree to complete the remainder of anti-TB treatment while in the study or
  * Had documented evidence of satisfactory anti-TB treatment as per WHO or national guidelines following review by a physician specializing in TB on entry to a qualifying study.
* Current or previous active TB regardless of treatment.
* Were temporarily discontinued from study intervention at the time of the final study visit of a qualifying study and, in the opinion of the investigator, participation in the extension study poses an unacceptable risk for the participant's participation.
* A new cancer or malignancy except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured by the investigator.
* Have developed any lymphoproliferative disorder during a qualifying study, such as Epstein Barr Virus (EBV) related lymphoproliferative disorder, or signs and symptoms suggestive of current lymphatic disease.
* Have significant uncontrolled cardiovascular, cerebrovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neuropsychiatric disorders, or abnormal laboratory values that developed during a qualifying study that, in the opinion of the investigator, poses an unacceptable risk for the participant's participation.
* Participants who are expected to be non-compliant with restrictions on medications and vaccinations prior to the study, during the study or during the 8-week safety follow-up of the study.
* Participants who are currently participating in any interventional clinical study other than a qualifying GSK3196165 clinical study.
* Abnormal chest radiograph within the last 12 weeks judged by the investigator as clinically-significant.
* Pregnant or lactating, or women planning to become pregnant or initiating breastfeeding.
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2916 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (267):
- United States (66):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Flagstaff, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Covina, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Palmetto Bay, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bowling Green, Kentucky
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Grand Blanc, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Freehold, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Minot, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Vandalia, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Yukon, Oklahoma
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Baytown, Texas
  - GSK Investigational Site, Colleyville, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Glendale, Wisconsin
- Argentina (16):
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Palta, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, San Isidro, Buenos Aires
  - GSK Investigational Site, San Nicolás de los Arroyos, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Nueva Cordoba
  - GSK Investigational Site, Salta
  - GSK Investigational Site, San Juan
- Australia (2):
  - GSK Investigational Site, Gold Coast, Queensland
  - GSK Investigational Site, Woodville, South Australia
- GSK Investigational Site, Mons, Belgium
- Bulgaria (7):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sevlievo
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Vidin
- Canada (2):
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Trois-Rivières, Quebec
- China (24):
  - GSK Investigational Site, Bengbu, Anhui
  - GSK Investigational Site, Guilin, Guangxi
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Zhuzhou, Hunan
  - GSK Investigational Site, Baotou, Inner Mongolia
  - GSK Investigational Site, Tongliao, Inner Mongolia
  - GSK Investigational Site, Taizhou, Jiangsu
  - GSK Investigational Site, Xuzhou, Jiangsu
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Pingxiang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Jinzhou, Liaoning
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Huzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Yangzhou
  - GSK Investigational Site, Yanji
- Colombia (3):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
- Czechia (6):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Praha 4 Nusle
  - GSK Investigational Site, Uherské Hradiště
  - GSK Investigational Site, Zlín
- Estonia (3):
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (4):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Rendsburg, Schleswig-Holstein
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Hungary (6):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szentes
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Veszprém
- India (10):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Belagavi
  - GSK Investigational Site, Hubli
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Surat
- Japan (21):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamaguchi
- Latvia (2):
  - GSK Investigational Site, Ādaži
  - GSK Investigational Site, Liepāja
- Lithuania (4):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Šiauliai
  - GSK Investigational Site, Vilnius
- Malaysia (4):
  - GSK Investigational Site, Klang
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Seremban, Negeri Sembilan
  - GSK Investigational Site, Sibu
- Mexico (8):
  - GSK Investigational Site, Mexicali, Baja California Sur
  - GSK Investigational Site, Mexico City, Durango
  - GSK Investigational Site, León, Guanajuato
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Durango
  - GSK Investigational Site, México
  - GSK Investigational Site, San Luis Potosí City
- Poland (21):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Grodzisk Mazowiecki
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Nowa Sól
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siedlce
  - GSK Investigational Site, Sochaczew
  - GSK Investigational Site, Staszów
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zamość
- Russia (14):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Korolyov
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tver'
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Belgrade, Serbia
- South Africa (10):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Bellville
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Kempton Park
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Stellenbosch
- South Korea (8):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Cheonan-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
- Spain (8):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela. La Coruña.
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Rajathevee
- Ukraine (11):
  - GSK Investigational Site, Cherkasy
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lutsk
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhzhia
  - GSK Investigational Site, Zaporizhzia
  - GSK Investigational Site, Zhytomyr
- United Kingdom (3):
  - GSK Investigational Site, Orpington, Kent
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Coventry

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Weinblatt ME, Taylor PC, McInnes IB, Atsumi T, Strand V, Takeuchi T, Bracher M, Brooks D, Curtis P, Gupta A, Nijhawan R, O'Shea C, Rayner K, Saurigny D, Shelton C, Wang M, Wang R, Fleischmann RM. Long-term safety and efficacy of anti-GM-CSF otilimab in patients with rheumatoid arthritis: long-term extension of three phase 3 randomised trials (contRAst X). BMJ Open. 2025 Mar 5;15(3):e088869. doi: 10.1136/bmjopen-2024-088869. PMID 40044198
- See also: 201790 contRAst 1 NCT03980483 — https://clinicaltrials.gov/ct2/show/NCT03980483?term=201790&draw=2&rank=2
- See also: 201791 contRAst 2 NCT03970837 — https://clinicaltrials.gov/ct2/show/NCT03970837?term=201791&draw=2&rank=2
- See also: 202018 contRAst 3 NCT04134728 — https://clinicaltrials.gov/ct2/show/NCT04134728?term=202018&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who consented, were enrolled and assigned to receive Otilimab 90 milligram (mg) or 150 mg weekly. Participants who received Otilimab in their qualifying study (202018, 201790 and 201791) were enrolled into this study on the same dose. Participants who received an active comparator in their qualifying study were centrally randomized using Interactive Response Technology (IRT) in a ratio of 1:1 to receive either Otilimab 90 mg or 150 mg weekly.
Pre-assignment Details: The participants in this study 209564 (ContRAst X) were adults with Rheumatoid Arthritis (RA) who completed the treatment phase of a qualifying Otilimab clinical study (Phase 3 studies 201790 [ContRAst 1], 201791 [ContRAst 2] or 202018 [ContRAst 3]) and who, in the investigator's and participant's judgement would have benefited from extended treatment with Otilimab. One participant withdrew from 150mg GSK3196165 before receiving intervention due to Physician Decision (N=1459).
Period: Overall Study
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Started | 1456 | 1459
Completed | 0 | 0
Not Completed | 1456 | 1459
Not completed — Adverse Event | 43 | 40
Not completed — Lack of Efficacy | 49 | 48
Not completed — Lost to Follow-up | 19 | 16
Not completed — Physician Decision | 17 | 20
Not completed — Withdrawal by Subject | 65 | 68
Not completed — INVESTIGATOR SITE CLOSED | 6 | 2
Not completed — PROTOCOL-SPECIFIED WITHDRAWAL CRITERION MET | 6 | 9
Not completed — STUDY TERMINATED BY SPONSOR | 1251 | 1256

BASELINE CHARACTERISTICS:
Population: One participant withdrew from 150mg GSK3196165 before receiving intervention due to Physician Decision. Hence the participant was removed from intent-to-treat (ITT) and safety population (N=1459).
Groups:
- Total: Total of all reporting groups
Arm/Group | Otilimab 90 mg | Otilimab 150 mg | Total
Number analyzed (Participants) | 1456 | 1459 | 2915
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 55.2 (11.38) | 55.7 (10.91) | 55.4 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1158 | 1181 | 2339
  Male | 298 | 278 | 576
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 40 | 53 | 93
  ASIAN | 223 | 206 | 429
  BLACK OR AFRICAN AMERICAN | 33 | 28 | 61
  WHITE | 1147 | 1157 | 2304
  MULTIPLE | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any untoward medical occurrence that, at any dose: results in death, cause life threatening events which requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly. Protocol defined AESIs were included.
Time Frame: Up to approximately 145 Weeks
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1456 | 1459
Participants
  Participants with AEs | 902 | 931
  Participants with SAEs | 123 | 114
  Participants with AESI | 120 | 95

2. Primary Outcome: Change From Baseline in Hematology Parameter of Platelet Count at Week 24
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter platelet count.
Time Frame: Baseline (Day 01) and Week 24
Population: The analysis was performed on the Safety Set that includes all randomized participants who received at least one dose of study treatment. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1180 | 1204
Giga cells per liter (10^9 cells/L) | -11.9 (66.86) | -9.7 (66.82)

3. Primary Outcome: Change From Baseline in Hematology Parameter of Platelet Count at Week 48
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter platelet count.
Time Frame: Baseline (Day 01) and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 706 | 702
Giga cells per liter (10^9 cells/L) | -12.5 (66.47) | -7.6 (71.36)

4. Primary Outcome: Change From Baseline in Hematology Parameter of Platelet Count at Week 96
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter platelet count.
Time Frame: Baseline (Day 01) and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 125 | 117
Giga cells per liter (10^9 cells/L) | -13.8 (60.72) | -5.7 (72.81)

5. Primary Outcome: Change From Baseline in Hematology Parameter of Platelet Count at Week 144
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter platelet count.
Time Frame: Baseline (Day 01) and Week 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1 | 2
Giga cells per liter (10^9 cells/L) | 17.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -37.5 (40.31)

6. Primary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter hemoglobin.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram Per Liter (g/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1195 | 1212
Gram Per Liter (g/L) | 0.4 (10.10) | 0.3 (9.89)

7. Primary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 48
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter hemoglobin.
Time Frame: Baseline (Day 01) and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram Per Liter (g/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 713 | 706
Gram Per Liter (g/L) | -0.5 (10.38) | -1.1 (10.62)

8. Primary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 96
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter hemoglobin.
Time Frame: Baseline (Day 01) and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram Per Liter (g/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 127 | 119
Gram Per Liter (g/L) | 1.0 (11.37) | 1.2 (10.24)

9. Primary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 144
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter hemoglobin.
Time Frame: Baseline (Day 01) and Week 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Gram Per Liter (g/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1 | 2
Gram Per Liter (g/L) | -1.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 2.0 (2.83)

10. Primary Outcome: Change From Baseline in White Blood Cell (WBC) Count With Differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils at Week 24
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including White Blood Cell (WBC) Count with Differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1350 | 1212
Giga cells per liter (10^9 cells/L)
  Neutrophils: number analyzed (Participants) | 1182 | 1208
  Neutrophils | -0.348 (2.18) | -0.390 (2.13)
  Lymphocytes: number analyzed (Participants) | 1182 | 1208
  Lymphocytes | -0.001 (0.55) | -0.012 (0.55)
  Monocytes: number analyzed (Participants) | 1182 | 1208
  Monocytes | 0.003 (0.18) | 0.00 (0.194)
  Eosinophils: number analyzed (Participants) | 1182 | 666
  Eosinophils | 0.027 (0.1623) | 0.022 (0.171)
  Basophils: number analyzed (Participants) | 1350 | 1208
  Basophils | -0.001 (0.0405) | -0.001 (0.04)
  Total WBC: number analyzed (Participants) | 1188 | 1212
  Total WBC | -0.32 (2.212) | -0.38 (2.230)

11. Primary Outcome: Change From Baseline in White Blood Cell (WBC) Count With Differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils at Week 48
Description: as for outcome 10
Time Frame: Baseline (Day 01) and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 709 | 703
Giga cells per liter (10^9 cells/L)
  Neutrophils: number analyzed (Participants) | 703 | 698
  Neutrophils | -0.318 (2.2215) | -0.541 (2.1426)
  Lymphocytes: number analyzed (Participants) | 703 | 698
  Lymphocytes | -0.022 (0.5385) | -0.051 (0.5725)
  Monocytes: number analyzed (Participants) | 703 | 698
  Monocytes | -0.002 (0.1871) | -0.013 (0.2461)
  Eosinophils: number analyzed (Participants) | 703 | 698
  Eosinophils | 0.018 (0.1435) | 0.028 (0.1844)
  Basophils: number analyzed (Participants) | 703 | 698
  Basophils | -0.004 (0.0391) | -0.006 (0.0403)
  Total WBC | -0.33 (2.283) | -0.58 (2.262)

12. Primary Outcome: Change From Baseline in White Blood Cell (WBC) Count With Differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils at Week 96
Description: as for outcome 10
Time Frame: Baseline (Day 01) and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 127 | 119
Giga cells per liter (10^9 cells/L)
  Neutrophils: number analyzed (Participants) | 127 | 44
  Neutrophils | -0.243 (1.8851) | -0.582 (2.4346)
  Lymphocytes: number analyzed (Participants) | 127 | 118
  Lymphocytes | 0.090 (0.6453) | 0.018 (0.5816)
  Monocytes: number analyzed (Participants) | 127 | 118
  Monocytes | -0.042 (0.2001) | -0.001 (0.2035)
  Eosinophils: number analyzed (Participants) | 127 | 118
  Eosinophils | 0.025 (0.1725) | 0.029 (0.1526)
  Basophils: number analyzed (Participants) | 127 | 118
  Basophils | -0.007 (0.0423) | -0.013 (0.0346)
  Total WBC | -0.18 (2.043) | -0.53 (2.568)

13. Primary Outcome: Change From Baseline in White Blood Cell (WBC) Count With Differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils at Week 144
Description: as for outcome 10
Time Frame: Baseline (Day 01) and Week 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1 | 2
Giga cells per liter (10^9 cells/L)
  Neutrophils | -0.360 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -0.935 (0.6718)
  Lymphocytes | -0.320 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 0.010 (0.3253)
  Monocytes | -0.220 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 0.010 (0.0424)
  Eosinophils: number analyzed (Participants) | 1 | 0
  Eosinophils | -0.130 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. |
  Basophils | 0.000 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 0.000 (0.0141)
  Total WBC | -1.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -0.85 (1.061)

14. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma Glutamyl Transferase (GGT), Creatine Kinase (CPK) at Week 24
Description: Blood samples were collected for the assessment of change from baseline in clinical chemistry parameters including AST, ALT, AP, GGT, CPK.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1232 | 1402
International units per liter (IU/L)
  Aspartate Aminotransferase (AST): number analyzed (Participants) | 1231 | 1242
  Aspartate Aminotransferase (AST) | 1.0 (11.09) | 0.8 (9.70)
  Alanine Aminotransferase (ALT): number analyzed (Participants) | 1232 | 1243
  Alanine Aminotransferase (ALT) | 0.0 (15.80) | -0.1 (15.20)
  Alkaline Phosphatase (AP): number analyzed (Participants) | 1232 | 1243
  Alkaline Phosphatase (AP) | 3.0 (18.85) | 3.1 (21.05)
  Gamma Glutamyl Transferase (GGT): number analyzed (Participants) | 1230 | 1402
  Gamma Glutamyl Transferase (GGT) | -0.9 (20.32) | -0.4 (18.94)
  Creatine Kinase (CPK): number analyzed (Participants) | 1230 | 1242
  Creatine Kinase (CPK) | 5.4 (103.03) | -3.8 (66.66)

15. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma Glutamyl Transferase (GGT), Creatine Kinase (CPK) at Week 48
Description: as for outcome 14
Time Frame: Baseline (Day 01) and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 762 | 749
International units per liter (IU/L)
  Aspartate Aminotransferase (AST): number analyzed (Participants) | 761 | 749
  Aspartate Aminotransferase (AST) | 0.4 (11.11) | 0.4 (11.32)
  Alanine Aminotransferase (ALT): number analyzed (Participants) | 762 | 748
  Alanine Aminotransferase (ALT) | -0.9 (16.35) | -1.2 (16.26)
  Alkaline Phosphatase (AP): number analyzed (Participants) | 762 | 748
  Alkaline Phosphatase (AP) | 5.4 (20.07) | 5.2 (21.32)
  Gamma Glutamyl Transferase (GGT): number analyzed (Participants) | 762 | 748
  Gamma Glutamyl Transferase (GGT) | -0.0 (22.44) | -0.4 (22.14)
  Creatine Kinase (CPK): number analyzed (Participants) | 762 | 748
  Creatine Kinase (CPK) | 7.8 (153.24) | -3.7 (71.52)

16. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma Glutamyl Transferase (GGT), Creatine Kinase (CPK) at Week 96
Description: as for outcome 14
Time Frame: Baseline (Day 01) and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 128 | 122
International units per liter (IU/L)
  Aspartate Aminotransferase (AST): number analyzed (Participants) | 128 | 44
  Aspartate Aminotransferase (AST) | 0.1 (11.65) | 2.0 (7.47)
  Alanine Aminotransferase (ALT): number analyzed (Participants) | 128 | 44
  Alanine Aminotransferase (ALT) | -2.4 (19.02) | -1.1 (9.33)
  Alkaline Phosphatase (AP): number analyzed (Participants) | 49 | 122
  Alkaline Phosphatase (AP) | 0.0 (18.98) | 8.6 (27.79)
  Gamma Glutamyl Transferase (GGT) | -1.9 (18.52) | -0.1 (19.67)
  Creatine Kinase (CPK) | 1.4 (39.73) | 3.6 (93.29)

17. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma Glutamyl Transferase (GGT), Creatine Kinase (CPK) at Week 144
Description: as for outcome 14
Time Frame: Baseline (Day 01) and Week 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1 | 2
International units per liter (IU/L)
  Aspartate Aminotransferase (AST) | -8.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 2.0 (0.0)
  Alanine Aminotransferase (ALT): number analyzed (Participants) | 1 | 0
  Alanine Aminotransferase (ALT) | -14.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. |
  Alkaline Phosphatase (AP) | 39.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -1.5 (6.36)
  Gamma Glutamyl Transferase (GGT) | -21.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 5.0 (14.14)
  Creatine Kinase (CPK) | -47.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -2.5 (31.82)

18. Primary Outcome: Change From Baseline in Lipid Profile Parameter of Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol, High-Density Lipoprotein-Cholesterol (HDL), Triglycerides at Week 24
Description: Blood samples was collected for the assessment of clinical chemistry parameters including Cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein-cholesterol (HDL), Triglycerides
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1183 | 1204
Millimoles per liter (mmol/L)
  Cholesterol: number analyzed (Participants) | 1183 | 1201
  Cholesterol | -0.038 (0.8542) | -0.011 (0.9685)
  HDL Cholesterol, Direct: number analyzed (Participants) | 1183 | 1201
  HDL Cholesterol, Direct | -0.020 (0.2703) | -0.022 (0.2869)
  LDL Cholesterol: number analyzed (Participants) | 1171 | 1190
  LDL Cholesterol | -0.031 (0.7239) | 0.010 (0.7818)
  Triglycerides | 0.033 (0.6503) | 0.011 (0.7895)

19. Primary Outcome: Change From Baseline in Lipid Profile Parameter of Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol, High-Density Lipoprotein-Cholesterol (HDL), Triglycerides at Week 48
Description: as for outcome 18
Time Frame: Baseline (Day 01) and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 730 | 719
Millimoles per liter (mmol/L)
  Cholesterol: number analyzed (Participants) | 730 | 718
  Cholesterol | -0.053 (0.9271) | -0.078 (0.9826)
  HDL Cholesterol, Direct: number analyzed (Participants) | 730 | 718
  HDL Cholesterol, Direct | -0.021 (0.2979) | -0.027 (0.2959)
  LDL Cholesterol: number analyzed (Participants) | 728 | 708
  LDL Cholesterol | -0.038 (0.7865) | -0.034 (0.7899)
  Triglycerides | 0.015 (0.6772) | -0.019 (0.7376)

20. Primary Outcome: Change From Baseline in Lipid Profile Parameter of Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol, High-Density Lipoprotein-Cholesterol (HDL), Triglycerides at Week 96
Description: as for outcome 18
Time Frame: Baseline (Day 01) and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 113 | 100
Millimoles per liter (mmol/L)
  Cholesterol | -0.178 (1.0350) | -0.130 (1.0570)
  HDL Cholesterol, Direct | -0.032 (0.2665) | -0.058 (0.3233)
  LDL Cholesterol: number analyzed (Participants) | 112 | 99
  LDL Cholesterol | -0.159 (0.8948) | -0.031 (0.8546)
  Triglycerides | 0.009 (0.8042) | -0.056 (0.7262)

21. Primary Outcome: Change From Baseline in Lipid Profile Parameter of Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol, High-Density Lipoprotein-Cholesterol (HDL), Triglycerides at Week 144
Description: as for outcome 18
Time Frame: Baseline (Day 01) and Week 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1 | 2
Millimoles per liter (mmol/L)
  Cholesterol | -2.360 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -2.240 (2.8709)
  HDL Cholesterol, Direct | 0.160 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -0.095 (0.0212)
  LDL Cholesterol | -2.250 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -1.750 (2.4183)
  Triglycerides | -0.580 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | -0.865 (0.9687)

22. Primary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE)>=Grade 3 Hematological/Clinical Chemistry Abnormalities
Description: Number of participants with NCI-CTCAE >=Grade 3 hematological/clinical chemistry abnormalities were summarized. Hematological and Clinical chemistry parameters were summarized according to the NCI-CTCAE, version 5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling. Higher grade indicates more severity. Data is presented for only those parameters for which participants had worst case >=Grade 3 shifts from Baseline.
Time Frame: Up to approximately 145 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1456 | 1459
Participants
  Hypercalcemia, Total, Grade 3 | 1 | 0
  Hyperkalemia, Total, Grade 4 | 2 | 0
  Hypernatremia, Total, Grade 3 | 1 | 0
  Hypernatremia, Total, Grade 4 | 0 | 1
  Chronic Kidney Disease, Total, Grade 3 | 0 | 1
  Creatinine increased, Total, Grade 3 | 1 | 0

23. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Total Score Lesser Than or Equal to (<=)10 (CDAI) Low Disease Activity (LDA) at Week 24, 48, 96 and 144
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Percentage values are rounded off.
Time Frame: Week 24, 48, 96 and 144
Population: The analysis was performed on the intent to treat (ITT) set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the subject was randomized to. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1206 | 1212
Percentage of participants
  Week 24 | 47.0 | 46.0
  Week 48: number analyzed (Participants) | 757 | 749
  Week 48 | 44.0 | 47.0
  Week 96: number analyzed (Participants) | 124 | 112
  Week 96 | 40.0 | 47.0
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 0.0

24. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Total Score <=2.8 (CDAI Remission) at Week 24, 48, 96 and 144
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8. Percentage values are rounded off.
Time Frame: Week 24, 48, 96 and 144
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the subject was randomized to. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1206 | 1212
Percentage of participants
  Week 24 | 11.0 | 10.0
  Week 48: number analyzed (Participants) | 757 | 749
  Week 48 | 12.0 | 9.0
  Week 96: number analyzed (Participants) | 124 | 112
  Week 96 | 13.0 | 9.0
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 0.0

25. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score Using 28 Joint Count and C-Reactive Protein (DAS28-CRP) <2.6 at Week 24, 48, 96 and 144
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). PtGA is transformed to a 0-10 scale before computing the total score. DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP greater than or equal to (<=)3.2. A negative change from baseline in DAS28-CRP indicates an improvement. Percentage values are rounded off.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1190 | 1199
Percentage of participants
  Week 24 | 26.0 | 25.0
  Week 48: number analyzed (Participants) | 719 | 715
  Week 48 | 25.0 | 25.0
  Week 96: number analyzed (Participants) | 108 | 99
  Week 96 | 26.0 | 28.0
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 0.0

26. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score Using 28 Joint Count and Erythrocyte Sedimentation Rate (ESR) <2.6 (DAS28-ESR Remission) at Week 24, 48, 96 and 132
Description: The DAS28-ESR is a measure of RA disease activity calculated using TJC28,SJC28, ESR (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). PtGA is transformed to a 0-10 scale before computing the total score. DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement. Percentage values are rounded off.
Time Frame: Week 24, 48, 96 and 132
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1084 | 1085
Percentage of participants
  Week 24 | 15.0 | 14.0
  Week 48: number analyzed (Participants) | 676 | 672
  Week 48 | 14.0 | 13.0
  Week 96: number analyzed (Participants) | 95 | 91
  Week 96 | 16.0 | 12.0
  Week 132: number analyzed (Participants) | 1 | 3
  Week 132 | 0.0 | 33.0

27. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) Remission at Week 24, 48, 96 and 144
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) <= 1, Swollen Joint Count 66 (SJC66) <= 1, high sensitivity C-reactive Protein (hsCRP) <= 1mg/dl and patient's global assessment of disease activity (PtGA) <= 10. Simple Disease Activity Index based ACR/EULAR remission is achieved if a has SDAI <= 3.3. The SDAI is the sum of the tender/painful joint count and swollen joint count, employing 28 joints; PtGA and PhGA (on a scale of 0-10); and hsCRP (mg/L). Percentage values are rounded off.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Number; unit: Percentage of participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1190 | 1199
Percentage of participants
  Boolean-based ACR/EULAR, Week 24 | 7.0 | 6.0
  Boolean-based ACR/EULAR, Week 48: number analyzed (Participants) | 719 | 715
  Boolean-based ACR/EULAR, Week 48 | 8.0 | 4.0
  Boolean-based ACR/EULAR, Week 96: number analyzed (Participants) | 108 | 99
  Boolean-based ACR/EULAR, Week 96 | 8.0 | 9.0
  Boolean-based ACR/EULAR, Week 144: number analyzed (Participants) | 0 | 1
  Boolean-based ACR/EULAR, Week 144 |  | 0.0

28. Secondary Outcome: Absolute Values for Clinical Disease Activity Index (CDAI) Total Score
Description: CDAI total score is a composite score consisting of the sum of TJC28, TJC28, PtGA (visual analogue scale with values from 0=best to 100=worst) and PhGA (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1206 | 1212
Scores on a scale
  Week 24 | 13.42 (10.669) | 14.26 (11.637)
  Week 48: number analyzed (Participants) | 757 | 749
  Week 48 | 13.85 (10.612) | 14.07 (11.186)
  Week 96: number analyzed (Participants) | 124 | 112
  Week 96 | 14.62 (11.443) | 15.22 (13.997)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 11.30 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

29. Secondary Outcome: Absolute Values for Disease Activity Score Using 28 Joint Count and C-Reactive Protein (DAS28-CRP)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- PtGA is transformed to a 0-10 scale before computing the total score. CRP scores range from 1.0 to 9.4, where lower scores indicate less disease activity.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1338 | 1199
Scores on a scale
  Week 24 | 3.49 (1.237) | 3.55 (1.269)
  Week 48: number analyzed (Participants) | 719 | 715
  Week 48 | 3.51 (1.224) | 3.54 (1.232)
  Week 96: number analyzed (Participants) | 108 | 99
  Week 96 | 3.44 (1.188) | 3.52 (1.389)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 3.21 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

30. Secondary Outcome: Absolute Values for Disease Activity Score Using 28 Joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). PtGA is transformed to a 0-10 scale before computing the total score. DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity.
Time Frame: Week 24, 48, 96 and 132
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1084 | 1085
Scores on a scale
  Week 24 | 3.97 (1.295) | 4.01 (1.333)
  Week 48: number analyzed (Participants) | 676 | 672
  Week 48 | 4.02 (1.284) | 4.05 (1.306)
  Week 96: number analyzed (Participants) | 95 | 91
  Week 96 | 3.92 (1.216) | 4.04 (1.470)
  Week 132: number analyzed (Participants) | 1 | 3
  Week 132 | 3.77 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 4.26 (1.560)

31. Secondary Outcome: Absolute Values of Van Der Heijde Modified Total Sharp Scores (mTSS)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score ranges from 0 to 448 for mTSS with higher values representing higher disease activity.
Time Frame: Week 24 and 48
Population: The analysis was performed on the ITT set that includes participants from qualifying studies 201790 and 201791 only who received at least one dose of study treatment. This population was based on the treatment the subject was randomized to. Number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 66 | 46
Scores on a scale
  Week 24 | 23.26 (34.191) | 30.31 (40.236)
  Week 48 | 23.27 (33.953) | 30.34 (40.432)

32. Secondary Outcome: Absolute Values for Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI includes 20 questions which assesses difficulty in performing activities of daily living. The questionnaire assesses eight domains of physical functioning: Dressing and Grooming, Hygiene, Arising, Reach, Eating, Grip, Walking, Common Daily Activities. The questions assess domain scores ranging from 0 "without any difficulty" to 3 "unable to do." Scores on each domain were summed and averaged to provide an overall score ranging from 0 to 3, where higher score reflected worse status and a lower score indicates better quality of life.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1228 | 1239
Scores on a scale
  Week 24 | 1.045 (0.6764) | 1.060 (0.6849)
  Week 48: number analyzed (Participants) | 768 | 764
  Week 48 | 1.072 (0.6679) | 1.096 (0.6691)
  Week 96: number analyzed (Participants) | 126 | 120
  Week 96 | 1.074 (0.6852) | 1.156 (0.7582)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 2.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

33. Secondary Outcome: Absolute Values for Arthritis Pain Visual Analogue Scale (VAS)
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1230 | 1239
Scores on a scale
  Week 24 | 34.6 (23.51) | 36.6 (23.85)
  Week 48: number analyzed (Participants) | 768 | 765
  Week 48 | 37.0 (23.55) | 36.0 (23.88)
  Week 96: number analyzed (Participants) | 127 | 119
  Week 96 | 39.3 (24.62) | 38.1 (27.08)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 26.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

34. Secondary Outcome: Absolute Values Short Form (SF)-36 Mental Component Scores (MCS)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health. Quality Metric software was used for scoring.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1228 | 1237
T-score
  Week 24 | 49.14 (10.386) | 49.44 (10.384)
  Week 48: number analyzed (Participants) | 768 | 764
  Week 48 | 49.54 (10.577) | 49.70 (10.557)
  Week 96: number analyzed (Participants) | 126 | 119
  Week 96 | 48.66 (11.483) | 49.75 (11.351)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 42.55 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

35. Secondary Outcome: Absolute Values SF-36 Domain Scores
Description: Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The MCS consists of 4 domains (social functioning, vitality, mental health, and role-emotional domains) and PCS consists of 4 domains (physical functioning, role-physical, bodily pain and general health). The individual question items are first summed for each item under the various sections. Then, those domain scores are weighted to a scale between 0 to 100, where higher score represents better health. Quality Metric software was used for scoring for SF-36.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1228 | 1237
Scores on a scale
  Bodily Pain at Week 24 | 54.49 (21.457) | 53.83 (21.158)
  Bodily Pain at Week 48: number analyzed (Participants) | 768 | 764
  Bodily Pain at Week 48 | 52.22 (21.099) | 52.94 (21.158)
  Bodily Pain at Week 96: number analyzed (Participants) | 126 | 119
  Bodily Pain at Week 96 | 49.90 (20.943) | 51.11 (21.983)
  Bodily Pain at Week 144: number analyzed (Participants) | 0 | 1
  Bodily Pain at Week 144 |  | 41.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  General Health at week 24 | 51.00 (18.744) | 50.30 (17.980)
  General Health at week 48: number analyzed (Participants) | 768 | 764
  General Health at week 48 | 50.35 (18.817) | 49.44 (17.645)
  General Health at week 96: number analyzed (Participants) | 216 | 119
  General Health at week 96 | 48.44 (20.029) | 46.73 (18.543)
  General Health at week 144: number analyzed (Participants) | 0 | 1
  General Health at week 144 |  | 45.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Mental Health at week 24 | 67.47 (19.387) | 68.05 (19.150)
  Mental Health at week 48: number analyzed (Participants) | 768 | 764
  Mental Health at week 48 | 67.64 (19.701) | 67.97 (19.636)
  Mental Health at week 96: number analyzed (Participants) | 126 | 119
  Mental Health at week 96 | 66.90 (20.860) | 68.49 (20.217)
  Mental Health at week 144: number analyzed (Participants) | 0 | 1
  Mental Health at week 144 |  | 50.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Physical Function at week 24 | 56.20 (25.644) | 55.28 (25.615)
  Physical Function at week 48: number analyzed (Participants) | 768 | 764
  Physical Function at week 48 | 54.23 (26.222) | 53.98 (25.397)
  Physical Function at week 96: number analyzed (Participants) | 126 | 119
  Physical Function at week 96 | 51.87 (25.735) | 50.92 (26.175)
  Physical Function at week 144: number analyzed (Participants) | 0 | 1
  Physical Function at week 144 |  | 35.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Role Emotional At week 24 | 74.79 (24.653) | 75.09 (24.760)
  Role Emotional At week 48: number analyzed (Participants) | 768 | 764
  Role Emotional At week 48 | 75.31 (24.008) | 76.18 (24.163)
  Role Emotional At week 96: number analyzed (Participants) | 126 | 119
  Role Emotional At week 96 | 73.35 (25.188) | 74.44 (26.324)
  Role Emotional At week 144: number analyzed (Participants) | 0 | 1
  Role Emotional At week 144 |  | 50.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Role Physical at week 24 | 58.58 (23.155) | 57.78 (23.514)
  Role Physical at week 48: number analyzed (Participants) | 768 | 764
  Role Physical at week 48 | 56.49 (23.645) | 57.57 (23.463)
  Role Physical at week 96: number analyzed (Participants) | 126 | 119
  Role Physical at week 96 | 54.27 (23.818) | 55.15 (24.956)
  Role Physical at week 144: number analyzed (Participants) | 0 | 1
  Role Physical at week 144 |  | 25.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Social Function at week 24 | 71.20 (24.001) | 71.39 (23.936)
  Social Function at week 48: number analyzed (Participants) | 768 | 764
  Social Function at week 48 | 70.88 (24.596) | 71.29 (24.123)
  Social Function at week 96: number analyzed (Participants) | 126 | 119
  Social Function at week 96 | 68.25 (24.065) | 69.43 (26.526)
  Social Function at week 144: number analyzed (Participants) | 0 | 1
  Social Function at week 144 |  | 62.50 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.
  Vitality at week 24 | 55.77 (20.690) | 55.18 (20.593)
  Vitality at week 48: number analyzed (Participants) | 768 | 764
  Vitality at week 48 | 55.24 (20.972) | 54.49 (21.262)
  Vitality at week 96: number analyzed (Participants) | 126 | 119
  Vitality at week 96 | 51.04 (23.127) | 54.25 (22.738)
  Vitality at week 144: number analyzed (Participants) | 0 | 1
  Vitality at week 144 |  | 50.00 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

36. Secondary Outcome: Absolute Values SF-36 Physical Component Scores (PCS)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health.PCS is primarily derived from 4 domains(PF,role-physical,BP,GH) representing overall physical health. Quality Metric software was used for scoring.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1228 | 1237
T-Score
  Week 24 | 41.19 (8.173) | 40.67 (8.232)
  Week 48: number analyzed (Participants) | 768 | 764
  Week 48 | 40.17 (8.586) | 40.13 (8.271)
  Week 96: number analyzed (Participants) | 126 | 119
  Week 96 | 39.18 (9.280) | 38.86 (8.879)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 35.03 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

37. Secondary Outcome: Absolute Values Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life.
Time Frame: Week 24, 48, 96 and 144
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1229 | 1238
Scores on a scale
  Week 24 | 36.0 (10.33) | 35.9 (10.25)
  Week 48: number analyzed (Participants) | 767 | 764
  Week 48 | 35.5 (10.53) | 35.4 (10.59)
  Week 96: number analyzed (Participants) | 126 | 119
  Week 96 | 35.2 (10.77) | 34.8 (11.87)
  Week 144: number analyzed (Participants) | 0 | 1
  Week 144 |  | 26.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived.

38. Secondary Outcome: Number of Participants With Anti-GSK3196165 Antibodies
Description: Serum samples were collected for the determination of anti- GSK3196165 antibodies (ADA) using a validated electrochemiluminescence (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Additionally, confirmed positive ADA samples were also tested in a validated neutralizing antibody assay to determine the potential neutralizing activity of the ADA
Time Frame: Week 120
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the subject was randomized to.
Measure: Count of Participants; unit: Participants
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1456 | 1459
Participants | 11 | 10

39. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Total Bilirubin, Direct Bilirubin at Week 24
Description: Blood samples were collected for the assessment of change from baseline in clinical chemistry parameters including total bilirubin, direct bilirubin.
Time Frame: Baseline (Day 01) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1232 | 1243
Micromoles per liter (umol/L)
  Total Bilirubin | 0.3 (2.87) | 0.3 (2.92)
  Direct Bilirubin: number analyzed (Participants) | 1224 | 1235
  Direct Bilirubin | 0.053 (0.764) | 0.027 (0.641)

40. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Total Bilirubin, Direct Bilirubin at Week 48
Description: as for outcome 39
Time Frame: Baseline (Day 01) and Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 762 | 749
Micromoles per liter (umol/L)
  Total Bilirubin | -0.0 (2.85) | 0.1 (3.04)
  Direct Bilirubin: number analyzed (Participants) | 757 | 743
  Direct Bilirubin | 0.011 (0.777) | 0.040 (0.690)

41. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Total Bilirubin, Direct Bilirubin at Week 96
Description: as for outcome 39
Time Frame: Baseline (Day 01) and Week 96
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 128 | 123
Micromoles per liter (umol/L)
  Total Bilirubin | -0.2 (3.22) | 0.5 (3.49)
  Direct Bilirubin: number analyzed (Participants) | 127 | 122
  Direct Bilirubin | 0.047 (0.815) | 0.041 (0.827)

42. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter Total Bilirubin, Direct Bilirubin at Week 144
Description: as for outcome 39
Time Frame: Baseline (Day 01) and Week 144
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
Number analyzed (Participants) | 1 | 2
Micromoles per liter (umol/L)
  Total Bilirubin | 4.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 4.5 (6.36)
  Direct Bilirubin | 2.000 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. | 1.500 (0.707)

ADVERSE EVENTS:
Time Frame: All AE and SAE were collected from the start of the study intervention. Initially the study was planned for 4 years approx. 208 weeks however due to early termination by sponsor; data for all Adverse event was collected up to approximately 145 Weeks only.
Arm/Group | Otilimab 90 mg | Otilimab 150 mg
All-Cause Mortality (participants affected / at risk) | 10/1456 | 9/1459
Serious Adverse Events (participants affected / at risk) | 123/1456 | 114/1459
Other Adverse Events (participants affected / at risk) | 279/1456 | 308/1459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otilimab 90 mg (N=1456) | Otilimab 150 mg (N=1459)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Omental haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 1 (2)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess bacterial (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 8 (8) | 10 (10)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 5 (5) | 5 (5)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0)
Viral sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Accidental poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (11)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 3 (3)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2) | 0 (0)
Device physical property issue (Product Issues) | 0 (0) | 1 (1)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Transient psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Brachiocephalic vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Otilimab 90 mg (N=1456) | Otilimab 150 mg (N=1459)
COVID-19 (Infections and infestations) | 141 (153) | 141 (148)
Upper respiratory tract infection (Infections and infestations) | 65 (74) | 88 (100)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 118 (158) | 129 (175)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT04333147/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT04333147/SAP_001.pdf